CLINICAL TRIAL: NCT01889810
Title: Effect of Vitamin D3 Supplementation on Insulin Resistance and Cardiovascular Risk Factors in People at High Risk of Type 2 Diabetes and Cardiovascular Disease (The DIR Study)
Brief Title: Effect of Vitamin D3 Supplementation on Insulin Resistance- The DIR Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Collaborators: Health and Social Care Research and Development , Northern Ireland (Other Government); Royal Victoria Hospital, Belfast (Other); Northern Ireland Chest Heart and Stroke (Other)
Responsible Party: Principal Investigator, Michelle McKinley, Senior Lecturer, Nutrition & Metabolism Research Group, Centre for Public Health, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: QUB: B12/35; HSC: 12117MMcK-AS
Record Dates: First submitted 2013-06-26; First posted 2013-06-28 (Estimated); Results first posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2022-06

CONDITIONS: Sub-optimal Vitamin D Status; Pre-diabetes; Insulin Resistance
Keywords: Vitamin D, Pre-diabetes, Insulin Resistance
MeSH Terms: conditions — Glucose Intolerance; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D3 supplementation (Active Comparator): Patients will take 3000IU (75 µg) Vitamin D3 supplementation per day for a period of 26 weeks.
  Interventions: Dietary Supplement: Vitamin D3 supplementation
- Placebo (Placebo Comparator): Placebo group
  Interventions: Dietary Supplement: Vitamin D3 supplementation

INTERVENTIONS:
Dietary Supplement: Vitamin D3 supplementation — 3000IU (75µg) vitamin D3 will be given daily for a period of 26 weeks to the group who receive the active comparator. The efficacy of vitamin D3 supplementation on insulin resistance will be compared to the placebo group.

SUMMARY:
Insulin resistance is a state where the body does not respond as it should to the insulin it produces. Individuals who are insulin resistant are at increased risk of both heart disease and type 2 diabetes; importantly, diabetes more than doubles the risk of heart disease, independent of other recognised risk factors. Interventions that prevent or reverse insulin resistance may help to attenuate risk of heart disease and diabetes. A number of randomised controlled trials provide proof of concept evidence regarding a beneficial effect of vitamin D on insulin resistance and other cardiovascular risk markers but experts have stated that further studies are required. Importantly, these studies should use appropriate endpoints, provide a high enough dose of vitamin D to optimise vitamin D status, and they should be conducted in clearly defined populations, The vitamin D trial we propose addresses these issues and aims to evaluate a potentially straightforward and low cost health care intervention for populations at highrisk of heart disease and diabetes. Specifically, this study would provide clinically relevant information on the metabolic effects of optimising vitamin D status in these high risk patients. This has clear economic and social implications given the current, and projected, burden of heart disease and diabetes.

This study will investigate the effect of vitamin D3 supplementation on insulin resistance and cardiovascular risk factors in people at high risk of type 2 diabetes and cardiovascular disease using the gold standard euglycaemic hyperinsulinaemic clamp method.

ELIGIBILITY:
Inclusion Criteria:

* Impaired glucose tolerance (Fasting glucose <7.0 mmol/L (126mg/dl) and 2hr post-glucose load 7.8-11.0 mmol/L (140-199 mg/dl) or Impaired fasting glucose 5.6-6.9 mmol/L (100-125mg/dL) defined according to American Diabetes Association
* Sub-optimal vitamin D status (<50nmol/L)

Exclusion Criteria:

* Diabetes mellitus
* Established cardiovascular disease
* Psychiatric problems
* Pregnant or lactating
* Medical conditions or dietary restrictions that would substantially limit ability to complete the study requirements
* Excessive alcohol consumption (>28 Units/week men or >21 Units/week women)
* Already taking vitamin D supplements > 10 µg/d
* Medical conditions or medications that could influence vitamin D metabolism
* History of kidney stones
* Hypercalcaemia
* Hyperparathyroidism
* Significant liver and renal disease (liver function tests >3x upper limit of normal and glomerular filtration rate <30ml/min)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2013-08; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle McKinley, PhD, Principal Investigator — Queen's University, Belfast
Locations (1):
- Queen's University, Belfast, Belfast, Northern Ireland, United Kingdom

REFERENCES:
- [Background] Wallace HJ, Holmes L, Ennis CN, Cardwell CR, Woodside JV, Young IS, Bell PM, Hunter SJ, McKinley MC. Effect of vitamin D3 supplementation on insulin resistance and beta-cell function in prediabetes: a double-blind, randomized, placebo-controlled trial. Am J Clin Nutr. 2019 Nov 1;110(5):1138-1147. doi: 10.1093/ajcn/nqz171. PMID 31559433

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vitamin D3 Supplementation | Placebo
Started | 35 | 31
Completed | 34 | 30
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin D3 Supplementation | Placebo | Total
Number analyzed (Participants) | 35 | 31 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (2.0) | 54.0 (1.7) | 53.3 (2.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 11 | 27
  Male | 19 | 20 | 39
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change in Insulin Resistance
Description: Insulin resistance will be measured using the gold standard euglycaemic-hyperinsulinaemic clamp method (note - it is anticipated that a total of 60 volunteers will complete the primary endpoint assessment).
Time Frame: Measured at baseline and after 6 months
Measure: Mean (Standard Deviation); unit: μmol/kg/min (Step 2 GIR corrected)
Arm/Group | Vitamin D3 Supplementation | Placebo
Number analyzed (Participants) | 33 | 29
μmol/kg/min (Step 2 GIR corrected) | 37.4 (13.8) | 36.3 (10.4)

2. Secondary Outcome: Change in Vitamin D Status
Description: Change in vitamin D status will be measured using the gold standard Ultra performance liquid chromatography followed by tandem mass spectrometry
Time Frame: Measured at baseline and after 6 months
Reporting Status: Not Posted

3. Secondary Outcome: Change in Markers of Cardiovascular Risk
Description: Measurements of seated and 24-hour ambulatory blood pressure, lipids, homeostasis model assessment (HOMA), HbA1c, and inflammatory and immune function markers including tumour necrosis factor-alpha and high sensitivity c-reactive protein
Time Frame: Measured at baseline and after 6 months
Reporting Status: Not Posted

4. Secondary Outcome: Change in Carotid-femoral Pulse Wave Velocity (PWV)
Description: Assessed by sequential tonometry with ECG gating using the SphygmoCor PWV System
Time Frame: Measured at baseline and after 6 months
Reporting Status: Not Posted

5. Secondary Outcome: Change in Hand Grip Strength
Description: Assessed using hand held dynamometer
Time Frame: Measured at baseline and after 6 months
Reporting Status: Not Posted

6. Secondary Outcome: Health Status
Description: SF-36 Questionnaire
Time Frame: Measured at baseline and after 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Vitamin D3 Supplementation | Placebo
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/31
Other Adverse Events (participants affected / at risk) | 0/35 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes